CLINICAL TRIAL: NCT03562910
Title: Pilot Study of a Novel Mobile-based Social Services Self-screening and Referral Tool in an Urban Pediatric Emergency Department
Brief Title: Mobile-based Social Services Screening and Referral Tool in an Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Verizon Foundation (Other)
Responsible Party: Principal Investigator, Amanda Stewart, Instructor of Pediatrics and Emergency Medicine, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P00026275
Record Dates: First submitted 2018-02-01; First posted 2018-06-20 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Poverty; Social Determinants of Health; Mobile Applications; Pediatric ALL; Emergencies
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All enrolled subjects will be given access to the HelpSteps application, either via their personal cell phone or to a provided tablet.
  Interventions: Other: HelpSteps application

INTERVENTIONS:
Other: HelpSteps application — Mobile or tablet-based tool that screens for social needs and refers to local agency based on needs and proximity.

SUMMARY:
This study will determine the feasibility and effectiveness of using a mobile-based social services screening and referral tool in an urban pediatric Emergency Department (ED). Families will be offered the option to either download the tool, known as HelpSteps, as a mobile application ("app") on a personal cell phone or to use the app on a provided tablet. After leading the family through a brief social needs screening survey, HelpSteps will recommend local social service agencies based on identified needs and location. Families will then complete a brief survey on the ease of use of the tool as well as receive a follow-up call to ask about usefulness of the tool in solving social problems. The investigators will also ask physicians to fill out a brief survey about the use of the tool in the ED.

DETAILED DESCRIPTION:
Many families presenting in the ED may have unmet social needs. Prior studies have shown that families are receptive to screening for these needs in the ED setting. HelpSteps is a screening tool that not only identifies social needs but also connects individuals with local health and social services agencies. There have been no studies to date assessing the use of a new mobile-version of HelpSteps or the use of the tool in the ED setting. The objective of this study is (1) to assess the feasibility of using a patient-centered social services screening and referral mobile tool in the ED and (2) to determine if the tool is useful in helping patients identify social needs and link to appropriate referral services post-ED visit.

Data will be collected in a prospective, non-randomized fashion using a convenience sample of 330 adult subjects. All parents will be screened for enrollment. If a parent is not present, all unaccompanied patients 18 and older will be screened instead. If there are both parents present, investigators will ask families to self-identify the most appropriate research subject by asking which parent in their family is typically responsible for household resources or applications. Non-English speaking families and patients who present with a triage score of 1 or 2 (high acuity) will be excluded.

Once enrolled, research subjects will be offered the option to either download HelpSteps on a personal cell phone or to use the application on a provided tablet. The subject will then open the Help Steps tool and complete a brief social needs screening survey. Based on the results of the screening and on geographic proximity, HelpSteps will recommend referral agencies personalized to the subject. The subject will then choose agencies they are interested in and receive a personalized list of referrals.

While still in the ED, families will be asked to complete a brief survey regarding ease of use and recommending the tool to family and friends. After the ED visit, subjects will be sent two electronic reminders asking if they would like a referral list resent. All participants will receive a follow-up phone call approximately 2 weeks post-study enrollment to ask whether they have used HelpSteps at home, whether or not they contacted a referral agency, if their social need(s) were resolved, and if the application was helpful in finding a solution to their need(s). The investigators will also ask physicians to fill out a brief survey about the impact of the tool on clinical flow and usefulness in help supplementing care for the patient.

The investigators plan to use descriptive statistics to evaluate three categories of data: (1) social services needs, referrals and follow-up, (2) usefulness of the HelpSteps application, and (3) physician perspectives on use of the HelpSteps in the ED. The investigators will analyze the mobile-based group and the tablet-based group separately as they are likely two different populations (based on the lower socioeconomic status and thus higher social needs associated with not having a phone).

ELIGIBILITY:
Inclusion Criteria:

* All parents/caregivers or patients 18 and older presenting to a pediatric emergency department

Exclusion Criteria:

* Non-English speaking
* Parents/caregivers or patients Families whose children are triaged to high acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of Social Needs | Day of enrollment
  Number of social needs categories screened positive for or selected as a need

SECONDARY OUTCOMES:
Number of referral agencies selected/contacted | Day of enrollment and Two weeks post-enrollment
  Participant selection and report of contacting social services organizations
Improvement in Social Needs | Two weeks post-enrollment
  Participant report of social need improved
Impact on clinical flow | Day of enrollment
  ED physician report of time added to encounter as a result of HelpSteps
ED physician attitudes towards social screening | Day of enrollment
  ED physician report on usefulness of HelpSteps

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Stewart, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bottino CJ, Rhodes ET, Kreatsoulas C, Cox JE, Fleegler EW. Food Insecurity Screening in Pediatric Primary Care: Can Offering Referrals Help Identify Families in Need? Acad Pediatr. 2017 Jul;17(5):497-503. doi: 10.1016/j.acap.2016.10.006. Epub 2017 Mar 13. PMID 28302365
- [Background] Fleegler EW, Lieu TA, Wise PH, Muret-Wagstaff S. Families' health-related social problems and missed referral opportunities. Pediatrics. 2007 Jun;119(6):e1332-41. doi: 10.1542/peds.2006-1505. PMID 17545363
- [Background] Hassan A, Scherer EA, Pikcilingis A, Krull E, McNickles L, Marmon G, Woods ER, Fleegler EW. Improving Social Determinants of Health: Effectiveness of a Web-Based Intervention. Am J Prev Med. 2015 Dec;49(6):822-31. doi: 10.1016/j.amepre.2015.04.023. Epub 2015 Jul 26. PMID 26215831